CLINICAL TRIAL: NCT05830955
Title: The Effect of Lullaby and Breastmilk Smell on Physiological Parameters, Comfort and Maternal Attachment Levels of Preterm Newborns
Brief Title: The Effect of Lullaby and Breastmilk Smell on Preterm Newborns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mustafa Kemal University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Yuzuncu Yil University (Other); Van Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gizem Kerimoğlu Yıldız, Assistant Professor, Mustafa Kemal University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: Hatay Mustafa Kemal University
Record Dates: First submitted 2023-03-15; First posted 2023-04-26 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Preterm; Infant, Premature, Diseases; Postpartum Depression; Mother-Infant Interaction
Keywords: Premature; Infant; Comfort; Maternal Attachment; Postpartum Depression
MeSH Terms: conditions — Premature Birth; Infant, Premature, Diseases; Depression, Postpartum | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be in three groups according to the interventions. The preterm newborns who are going to listen a live lullaby from their mothers' voice will be the first group (Lullaby group). The preterms in the second group (Breast milk group) are going to smell their mothers' breast milk. The preterms in the third group (Control group) are going to recieve rutin nursing care interventions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lullaby Group (Experimental): The preterm newborns who are going to listen a live lullaby from their mothers' voice will be the first group (Lullaby group).
  Interventions: Other: Lullaby group
- Breast milk Group (Experimental): The preterms in the second group (Breast milk group) are going to smell their mothers' breast milk.
  Interventions: Other: Breast milk group
- Control Group (Other): The preterms in the third group (Control group) are going to recieve rutin nursing care interventions.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Lullaby group — The preterm newborns who are going to listen a live lullaby from their mothers' voice will be the first group (Lullaby group).
  Arms: Lullaby Group
Other: Breast milk group — The preterms in the second group (Breast milk group) are going to smell their mothers' breast milk.
  Arms: Breast milk Group
Other: Control group — The preterms in the third group (Control group) are going to recieve rutin nursing care interventions.
  Arms: Control Group

SUMMARY:
The goal of this clinical trial is to investigate the effect of live lullaby from mother voice, and breast milk smell on pyhsiological parameters, comfort and maternal attachment levels of preterm newborns who are between 35-37 weeks of gestation at the time of the study and the level of pospartum depression of mothers. The main hypothesis are:

H0: The live lullaby from mother voice and breast milk smell have no effects on pyhsiological parameters, comfort and maternal attachment levels of preterm newborns H1: The live lullaby from mother voice has effects on pyhsiological parameters, comfort and maternal attachment levels of preterm newborns H2: The breast milk smell has effects on pyhsiological parameters, comfort and maternal attachment levels of preterm newborns H3: There is differences between the live lullaby from mother voice and the breast milk smell interventions in terms of preterm newborns' physiological parameters, comfort and maternal attachment levels.

H4: The postpartum depression level of mothers in experimental groups (lullaby group and breast milk group) is lower than the control group.

Participants will be in three groups according to the interventions. The preterm newborns who are going to listen a live lullaby from their mothers' voice will be the first group (Lullaby group). The preterms in the second group (Breast milk group) are going to smell their mothers' breast milk. The preterms in the third group (Control group) are going to recieve rutin nursing care interventions.

ELIGIBILITY:
Inclusion Criteria:

* Parents' willingness to participate in the study
* Turkish literate parents
* Babies between 35-37 weeks of gestation
* Apgar score of 7 or higher at birth
* Stability of the baby (near discharge)
* Having mother's milk

Exclusion Criteria:

* Parents' reluctance to participate in the study
* Babies younger than 35 weeks and older than 37 weeks
* Babies receiving phototherapy
* Finding a congenital anomaly in infants
* Apgar score below 7 at birth
* Being connected to a mechanical ventilator

Ages: 35 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 57 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-03-04 (Actual); Study Completion 2024-03-05 (Actual)

PRIMARY OUTCOMES:
Heart Rate change | 5 minutes before the intervention, during the intervention (5th and 10th minutes) and 5 minutes after the application, for 3 consecutive days.
  Heart Rate change before, during and after the intervention
Oxygen Saturation change | 5 minutes before the intervention, during the intervention (5th and 10th minutes) and 5 minutes after the application, for 3 consecutive days.
  Oxygen Saturation change before, during and after the intervention
Respiration Rate change | 5 minutes before the intervention, during the intervention (5th and 10th minutes) and 5 minutes after the application, for 3 consecutive days.
  Respiration Rate change before, during and after the intervention
Body Temperature change | 5 minutes before the intervention, during the intervention (5th and 10th minutes) and 5 minutes after the application, for 3 consecutive days.
  Body Temperature change before, during and after the intervention
Comfort level change | 5 minutes before the intervention, during the intervention (5th and 10th minutes) and 5 minutes after the application, for 3 consecutive days
  Premature Infant Comfort Behavior Scale (ComfortNeo) will be used before, during and after the intervention. Each item of this five-point Likert scale is scored from 1 to 5 from bad to good. The baby's comfort is evaluated according to the total score. Accordingly, 30 indicates the lowest and 6 the highest comfort score. A high score on the scale indicates a low level of comfort.
Maternal Attachment | 28 days after discharge
  Maternal Attachment Scale This scale consists of 26 items and is in 4-point Likert type. "Always" is calculated as 4 points, "often" as 3 points, "sometimes" as 2 points, and "never" as 1 point. An overall score is obtained from the sum of all items. The lowest score to be obtained from the scale is 26, and the highest score is 104. A high score indicates high maternal attachment.
Postpartum Depression | Before the interventions and 28 days after discharge
  Edinburgh Postpartum Depression Scale The scale is in the form of a four-point Likert scale and consists of a total of 10 items. Items 1,2 and 4 are scored as 0,1,2,3 and other items as 3,2,1.0. The lowest possible score is 0 and the highest score is 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Training and Research Hospital, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The researchers have not planned to share any individual participant data yet.

REFERENCES:
- [Background] Rattaz C, Goubet N, Bullinger A. The calming effect of a familiar odor on full-term newborns. J Dev Behav Pediatr. 2005 Apr;26(2):86-92. doi: 10.1097/00004703-200504000-00003. PMID 15827459
- [Background] Namjoo R, Mehdipour-Rabori R, Bagherian B, Nematollahi M. Comparing the effectiveness of mother's live lullaby and recorded lullaby on physiological responses and sleep of preterm infants: a clinical trial study. J Complement Integr Med. 2021 May 24;19(1):121-129. doi: 10.1515/jcim-2020-0507. PMID 34022122
- [Background] Cignacco E, Hamers JP, van Lingen RA, Zimmermann LJ, Muller R, Gessler P, Nelle M. Pain relief in ventilated preterms during endotracheal suctioning: a randomized controlled trial. Swiss Med Wkly. 2008 Nov 1;138(43-44):635-45. doi: 10.4414/smw.2008.12288. PMID 19005869
- [Background] Lessen Knoll BS, Daramas T, Drake V. Randomized Controlled Trial of a Prefeeding Oral Motor Therapy and Its Effect on Feeding Improvement in a Thai NICU. J Obstet Gynecol Neonatal Nurs. 2019 Mar;48(2):176-188. doi: 10.1016/j.jogn.2019.01.003. Epub 2019 Feb 2. PMID 30721652
- [Background] da Silva CM, Cacao JM, Silva KC, Marques CF, Merey LS. Physiological responses of preterm newborn infants submitted to classical music therapy. Rev Paul Pediatr. 2013 Jan-Mar;31(1):30-6. doi: 10.1590/s0103-05822013000100006. English, Portuguese. PMID 23703041
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Aydin N, Inandi T, Yigit A, Hodoglugil NN. Validation of the Turkish version of the Edinburgh Postnatal Depression Scale among women within their first postpartum year. Soc Psychiatry Psychiatr Epidemiol. 2004 Jun;39(6):483-6. doi: 10.1007/s00127-004-0770-4. PMID 15205733
- [Background] Kurt FY, Kucukoglu S, Ozdemir AA, Ozcan Z. The effect of kangaroo care on maternal attachment in preterm infants. Niger J Clin Pract. 2020 Jan;23(1):26-32. doi: 10.4103/njcp.njcp_143_18. PMID 31929203
- [Background] Loewy J, Stewart K, Dassler AM, Telsey A, Homel P. The effects of music therapy on vital signs, feeding, and sleep in premature infants. Pediatrics. 2013 May;131(5):902-18. doi: 10.1542/peds.2012-1367. Epub 2013 Apr 15. PMID 23589814
- [Background] Alipour Z, Eskandari N, Ahmari Tehran H, Eshagh Hossaini SK, Sangi S. Effects of music on physiological and behavioral responses of premature infants: a randomized controlled trial. Complement Ther Clin Pract. 2013 Aug;19(3):128-32. doi: 10.1016/j.ctcp.2013.02.007. Epub 2013 May 9. PMID 23890458
- [Background] Taheri L, Jahromi MK, Abbasi M, Hojat M. Effect of recorded male lullaby on physiologic response of neonates in NICU. Appl Nurs Res. 2017 Feb;33:127-130. doi: 10.1016/j.apnr.2016.11.003. Epub 2016 Nov 9. PMID 28096005